CLINICAL TRIAL: NCT03105908
Title: Internet-delivered ACT Treatment for Patients With Chronic Pain: A Randomized Controlled Trial
Brief Title: Internet-delivered ACT for Chronic Pain
Acronym: iACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rikard Wicksell (Other)
Collaborators: AFA Insurance (Industry)
Responsible Party: Sponsor-Investigator, Rikard Wicksell, Director of Functional Area Medical Psychology, Karolinska Univ Hospital, assoc professor and head of research group Behavior Medcine, Karolinska Institutet, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015/1638-31/2
Record Dates: First submitted 2017-03-15; First posted 2017-04-10 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Other): Internet delivered Acceptance and Commitment therapy, supported by a psychologist/psychology student under supervision.
  Interventions: Behavioral: Internet delivered Acceptance and Commitment therapy
- Waiting list control condition (Other): Participants receive no treatment for ten weeks, i.e. waiting list condition. Following post-assessment, the control condition receive unguided iACT (i.e. the same content and structure as iACT but without systematic therapist communication).
  Interventions: Behavioral: Waiting list control condition

INTERVENTIONS:
Behavioral: Internet delivered Acceptance and Commitment therapy — The main component in the treatment is exposure to symptoms and feared situations. The iACT program is adapted from the evidence based face-to-face treatment at the Behavioral Medicine unit at Karolinska University Hospital. The iACT program has a different structure but is equal in content to face-to-face treatment, and is to be completed within ten weeks. Participants receive texts, audio files, movies and exercises and have online contact with their psychologist via an internet platform or a smart phone application. The treatment aims to encourage valued behaviors in the presence of inner discomfort.
  Other Names: iACT
  Arms: Treatment
Behavioral: Waiting list control condition — After a ten week wait list period, the control condition receive same treatment as the intervention group, but without therapist support.
  Arms: Waiting list control condition

SUMMARY:
The overall aim of the present study is to evaluate an internet-delivered Acceptance and Commitment therapy treatment (iACT) for patients with chronic pain. More specifically, the study will evaluate if 1) iACT is effective in improving functioning and quality of life in comparison to a waitlist condition, 2) if iACT is cost-effective, 3) factors that influence treatment outcome (i.e. predictors, moderators or characteristics of treatment responders), 4) if psychological variables mediates the effects of treatment on outcome, and 5) if subgroups of patients varies in change processes (i.e. moderated mediation).

The main hypothesis is that iACT will improve functioning and quality of life.

DETAILED DESCRIPTION:
Chronic pain affects 12-30% of the population and often results in depression, disability, and reduced quality of life. Medical strategies are often ineffective or insufficient to alleviate symptoms and increase functioning. Instead, the empirical support for cognitive behavior therapy (CBT) is today well established, and such interventions are commonly seen as critically important for patients with chronic pain. However, modest effects sizes calls for further improvements. Recent developments within CBT, particularly Acceptance and Commitment Therapy (ACT), have suggested the utility of acceptance and mindfulness strategies to manage pain and distress. The body of evidence for ACT has grown rapidly during the past decade, and ACT is today listed by the American Psychological Association as a treatment for chronic pain, with strong empirical support.

Internet-delivered ACT

Despite the increased empirical support for ACT the availability is still very limited, and a large number of patients do not receive this treatment. In other domains, the accessibility of empirically supported treatments has increased during the past decade due to the development of methods to deliver the treatment via internet. For example, a large number of studies illustrate the utility of internet-delivered CBT for anxiety, insomnia and depression, with treatment effects similar to those obtained in studies with face-to-face treatment. Few studies have yet evaluated internet-delivered ACT (iACT) for chronic pain, but a recent pilot study from our group with participants suffering from fibromyalgia (n=41) illustrated very promising results that warrant further studies to evaluate the effects of this treatment.

Moderators and mediators of treatment outcome

If iACT shows to be effective, it is vital to identify for whom this treatment works. For example, it is possible that factors such as age, pain duration or depression may moderate the effects of treatment. Also, it is likely that some individuals who respond well to regular face-to-face treatment do not benefit from internet-delivered interventions. Furthermore, recent studies have shown that acceptance of pain and distress may be a more important mediator of change than e.g. pain intensity, catastrophizing or anxiety. However, no study has to our knowledge yet explored if subgroups of patients (e.g. men and women) improve via different change processes (i.e. moderated mediation). More information regarding moderators and mediators of change will make it possible to adjust and tailor interventions to meet specific individual needs, and thereby increase the effects of treatment.

Recruitment

Patients will be recruited through self referral. Thus, information regarding the study will be provided through newspapers and social media, as well as in direct communication with pain clinics and primary care units, including instructions regarding e.g. eligibility and how to sign up. Once patients have been found eligible and expressed interest in study participation they will be assessed by a psychologist, and when needed by a pain physician, via semi-structured interviews to confirm eligibility and to ensure that the patient meet the study criteria. Informed consent is obtained from all participants prior to the assessment.

Statistical methods

Evaluations of treatment effects are primarily based on intent-to-treat analyses. The statistical approach will primarily be based on linear multilevel modeling (LMM), which takes into account dependencies between repeated measures and differences between patients in pre-treatment status and treatment response (i.e. random effects modeling) and also provide means of handling missing data. More traditional methods, such as ANOVA and hierarchical regression, may also be utilized when appropriate. Analyses of change processes (mediation, moderation, moderated mediation) will follow guidelines and recommendations (e.g. cross-product of coefficients approach, bootstrapping). The main health economic outcomes will be the incremental cost-effectiveness ratio, which is a measure of the relationship between the cost of the treatment and the incremental value it provides in terms of functioning, compared to the control condition.

ELIGIBILITY:
Inclusion Criteria:

* a pain duration of ≥ 6 months;
* are able to communicate in Swedish
* have access to computer and internet in their home environment.
* have access to a cell phone with the possibility of receiving text messages
* no planned changes in medication use, or any other changes in interventions for their pain planned

Exclusion Criteria:

* injury or illness that require immediate assessment or different treatment, or that is expected to progress significantly during the next 6 months
* unstable medication (planned changes in medication during next 4 months)
* previous ACT or CBT treatment during the past 3 months
* severe psychiatric co-morbidity (e.g. high risk of suicide) as assessed by the psychologist in a semi-structured interview

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2017-03-16 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Pain Interference Index (changes between assessments) | Baseline, 10 weekly ratings, post (10 weeks), follow ups three, six and twelve months post treatment
  Self rated measure of daily functioning related to pain

SECONDARY OUTCOMES:
The Valuing Questionnaire (changes) | Baseline, mid (4 weeks), post (10 weeks), follow ups three, six and twelve months post treatment
  Self rated progress and obstacles in valued actions
Psychological Inflexibility in Pain Scale (changes) | Baseline, 10 weekly ratings, post (10 weeks), follow ups three, six and twelve months post treatment
  Self rated psychological inflexibility related to pain
Patient Health Questionnaire 9 (changes) | Baseline, post (10 weeks), follow ups three, six and twelve months post treatment
  Self rated depressive symptoms
European Quality of Life Five Dimensions Questionnaire (changes) | Baseline, post (10 weeks), follow ups three, six and twelve months post treatment
  Self rated quality of life
Insomnia Severity Index (changes) | Baseline, post (10 weeks), follow ups three, six and twelve months post treatment
  Self rated degree of insomnia
Pain Intensity (changes) | Baseline, post (10 weeks), follow ups three, six and twelve months post treatment
  Self rated degree of pain during the last week on a scale from 0-10
Occupational status (changes) | Baseline, post (10 weeks), follow ups three, six and twelve months post treatment
  Self reported occupational status indicated on a pre specified list, including sick leave and/or retirement
Perceived Stress Scale - 4 items (changes) | Baseline, post (10 weeks), follow ups three, six and twelve months post treatment
  Self rated level of perceived stress
General Anxiety Disorder - 7 item (changes) | Baseline, post (10 weeks), follow ups three, six and twelve months post treatment
  Self rated symptoms of general anxiety
Medication use (changes) | Baseline, post (10 weeks), follow ups three, six and twelve months post treatment
  Self reported medicine use

CONTACTS AND LOCATIONS:
Overall Officials: Rikard Wicksell, PhD, MSc, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gentili C, Zetterqvist V, Rickardsson J, Holmstrom L, Ljotsson B, Wicksell R. Examining predictors of treatment effect in digital Acceptance and Commitment Therapy for chronic pain. Cogn Behav Ther. 2023 Jul;52(4):380-396. doi: 10.1080/16506073.2023.2191826. Epub 2023 Mar 27. PMID 36971108